CLINICAL TRIAL: NCT04860765
Title: Congenital Multicenter Trial of Pulmonic Valve Dysfunction Studying the SAPIEN 3 Interventional THV Post-Approval Study
Brief Title: COMPASSION S3 Post-Approval Study
Status: Active, not recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-07
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Complex Congenital Heart Defect; Dysfunctional RVOT Conduit; Pulmonary Valve Insufficiency; Pulmonary Valve Degeneration; Pulmonary Valve; Obstruction
Keywords: Transcatheter pulmonary valve replacement; Transcatheter pulmonary valve implantation; SAPIEN 3
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: US Export: No

GROUPS / COHORTS (1):
- TPVR: Subjects with a dysfunctional RVOT conduit or previously implanted surgical valve in the pulmonic position will undergo transcatheter pulmonary valve replacement (TPVR).
  Interventions: Device: SAPIEN 3 THV

INTERVENTIONS:
Device: SAPIEN 3 THV — SAPIEN 3 THV in the pulmonic position

SUMMARY:
This study will monitor device performance and outcomes of the SAPIEN 3 Transcatheter Heart Valve (THV) System in subjects with a dysfunctional right ventricular outflow tract (RVOT) conduit or previously implanted surgical valve in the pulmonic position with a clinical indication for intervention.

DETAILED DESCRIPTION:
This is a single arm, prospective, multicenter post-approval study.

ELIGIBILITY:
Inclusion Criteria:

1. Dysfunctional RVOT conduit or previously implanted surgical valve
2. RVOT/PV with ≥ moderate regurgitation and/or a mean RVOT/PV gradient of ≥ 35 mmHg

Exclusion Criteria:

1. Inability to tolerate an anticoagulation/antiplatelet regimen
2. Active bacterial endocarditis or other active infections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with a dysfunctional RVOT conduit or previously implanted surgical valve in the pulmonic position with a clinical indication for intervention
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Device Success | Discharge, expected to be within 1-5 days post-procedure
  Defined as a composite of:
  * Single THV implanted in the desired location
  * Right ventricle to pulmonary artery peak-to-peak gradient < 35 mmHg post-implantation
  * Less than moderate PR by discharge TTE
  * Free of explant at 24 hours post-implantation

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - Cedars Sinai, Los Angeles, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Advocate Childrens Hospital, Oak Lawn, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Minneapolis Heart, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Mount Sinai, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinatti Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Dell Children's, Austin, Texas
  - Children's Health Dallas, Dallas, Texas
  - Primary Children's, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No